CLINICAL TRIAL: NCT01817673
Title: Creatine Supplementation on Kidney Function in Resistance-trained Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: Creatine & kidney
Record Dates: First submitted 2013-03-20; First posted 2013-03-25 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-03

CONDITIONS: Healthy Persons
MeSH Terms: interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- creatine (Experimental): 20 g/d for 5 d followed by 5 g/d throughout the trial
  Interventions: Dietary Supplement: creatine
- placebo (dextrose) (Placebo Comparator): 20 g/d for 5 d followed by 5 g/d throughout the trial
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: creatine — 20 g/d for 5 d followed by 5 g/d throughout the trial
  Arms: creatine
Dietary Supplement: placebo
  Arms: placebo (dextrose)

SUMMARY:
There is a claim that creatine supplementation might affect kidney function, especially in those consuming a high-protein diet. The aim of this study was to investigate the effects of creatine supplementation on kidney function in resistance-trained individuals ingesting a high-protein diet.

ELIGIBILITY:
Inclusion Criteria:

* participation in recreational resistance training
* consumption of a high-protein diet (≥ 1.2 g/Kg/d)

Exclusion Criteria:

* vegetarian diet
* use of creatine supplements in the past 6 months
* chronic kidney disease
* use of anabolic steroids.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2011-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
kidney function | 3 months
  as assessed by 51Cr-EDTA clearance

SECONDARY OUTCOMES:
proteinuria | 3 months
albuminuria | 3 months
serum urea | 3 months
serum creatinine | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Gualano, Professor, Principal Investigator — University of Sao Paulo
Locations (1):
- Univsersity of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Lugaresi R, Leme M, de Salles Painelli V, Murai IH, Roschel H, Sapienza MT, Lancha Junior AH, Gualano B. Does long-term creatine supplementation impair kidney function in resistance-trained individuals consuming a high-protein diet? J Int Soc Sports Nutr. 2013 May 16;10(1):26. doi: 10.1186/1550-2783-10-26. PMID 23680457